CLINICAL TRIAL: NCT01858077
Title: Amsterdam Investigator-initiateD Absorb Strategy All-comers Trial (AIDA Trial): A Clinical Evaluation Comparing the Efficacy and Performance of ABSORB™ Everolimus Eluting Bioresorbable Vascular Scaffold Strategy Versus the XIENCE Family (XIENCE PRIME™ or XIENCE Xpedition™) Everolimus Eluting Coronary Stent Strategy in the Treatment of Coronary Lesions in Consecutive All-comers.
Brief Title: Amsterdam Investigator-initiateD Absorb Strategy All-comers Trial
Acronym: AIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.J. Wykrzykowska, J.J. Wykrzykowska, MD, PhD, Coordinating Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COR 10341; AIDA trial (Registry Identifier: AIDA trial)
Record Dates: First submitted 2013-05-10; First posted 2013-05-21 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABSORB BVS™ (Active Comparator): Abbott Vascular ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold System
  Interventions: Device: ABSORB BVS™
- XIENCE™ (Active Comparator): XIENCE PRIME everolimus eluting coronary stent system and the XIENCE Xpedition everolimus eluting coronary stent system
  Interventions: Device: XIENCE™

INTERVENTIONS:
Device: ABSORB BVS™ — Bioresorbable scaffold
  Other Names: ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold; ABSORB; ABSORB BVS; BVS
  Arms: ABSORB BVS™
Device: XIENCE™ — Drug eluting metallic stent
  Other Names: XIENCE PRIME; XIENCE Xpedition; XIENCE; DES; Drug eluting stent
  Arms: XIENCE™

SUMMARY:
To evaluate the efficacy and performance in an all-comers contemporary population of the ABSORB bioresorbable vascular scaffolds (BVS) strategy versus the XIENCE family (XIENCE PRIME or XIENCE Xpedition) everolimus eluting coronary stent system in the treatment of coronary lesions.

DETAILED DESCRIPTION:
The AIDA trial is a prospective, randomized (1:1), active control, single blinded, four-center, all-comers, non-inferiority trial. A total of 1845 patients were enrolled. The study population includes both simple and complex lesions, as well as stable and acute coronary syndrome patients. The follow-up will continue for 5 years including clinical endpoint characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions and the Instructions for Use of the ABSORB BVS strategy and XIENCE family.
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the ABSORB BVS strategy and he/she or his/her legally authorized representative provides written informed consent prior to any Clinical Investigation related procedure, as approved by the appropriate Ethics Committee.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject has a true bifurcation lesion where a priori two scaffold/stent strategy is planned.
* Unsuccessful predilation of one or more of the planned lesion to be treated.
* Planned treatment of in-stent restenosis of a previously placed metallic stent.
* Subject has one or more lesion planned to be treated with a scaffold/stent diameter size smaller than 2.5 mm or greater than 4.0 mm.
* Subject has one or more lesion planned to be treated with a stent/scaffold length greater than 70 mm and/or overlapping of four or more scaffolds/stents.
* Subject has known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel, prasugrel and ticagrelor, inclusive), everolimus, poly (L-lactide), poly (DL-lactide), cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
* Subjects pregnant or nursing subjects and those who plan pregnancy in the period up to 2 years following index procedure. (Female subjects of child-bearing potential must have a negative pregnancy test done within 28 days prior to the index procedure and contraception must be used during participation in this trial)
* Subjects with a limited life expectancy less than one year.
* Subjects with factors that impede clinical follow-up (e.g. no fixed abode).
* Subject is already participating in another clinical investigation that has not yet reached its primary endpoint.
* Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff or sponsor staff) or subject unable to read or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1845 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 2 years
  The primary composite endpoint is the device-oriented composite of target vessel failure (TVF):
  * Cardiac death
  * Myocardial Infarction (MI) (unless clearly attributable to a non target vessel)
  * Target vessel revascularization

SECONDARY OUTCOMES:
Device success | 1 day
  Successful delivery and deployment of the first study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 20% by quantitative coronary angiography (QCA) and thrombolysis in myocardial infarction (TIMI) 3 flow grade of the treated vessel.
Procedural success | 1 day
  Achievement of final in-scaffold/stent residual stenosis of less than 20% by QCA and TIMI 3 flow grade of the treated vessel with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat Target Lesion Revascularization during the hospital stay.
Target vessel failure (TVF) | 30 days, and 1, 3, 4 and 5 years
  Cardiac death, MI (not clearly attributable to a nontarget vessel) or target vessel revascularization
Target lesion failure | 30 days, and 1, 2, 3, 4 and 5 years
  Cardiac death, MI (not clearly attributable to a nontarget vessel) or target lesion revascularization
All revascularizations | 5 year
Major adverse cardiac events | 30 days, and 1, 2, 3, 4 and 5 years
  All-cause mortality, any MI, any repeat revascularization
All cause mortality | 30 days, 1 year, 2, 3, 4 and 5 years
Myocardial Infarction | 30 days, 1, 2, 3, 4 and 5 years
  Q-wave Myocardial Infarction (QMI) and non Q-wave Myocardial Infarction (nonQMI)/target-vessel myocardial infarction (TVMI) and non-TVMI
Target Lesion Revascularization (TLR) | 30 days, 1 year, 2, 3, 4 and 5 years
Target Vessel Revascularization (TVR) | 30 days, 1 year, 2, 3, 4 and 5 years
Non-Target Vessel Revascularization (NTVR) | 30 days, 1 year, 2, 3, 4 and 5 years
Scaffold/Stent Thrombosis | 30 days, 1, 2, 3, 4 and 5 years
  acute, subacute, late/definite and probable
Seattle Angina Questionnaire (SAQ) | 1 year and 2 years
Quality of Life Questionnaire (QOL) | 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Wykrzykowska, MD, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Rob de Winter, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jan Piek, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jan Tijssen, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jose Henriques, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (5):
- Netherlands (5):
  - AMC, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - TerGooi Hospital, Hilversum
  - Medical Center Leeuwarden, Leeuwarden

REFERENCES:
- [Background] Woudstra P, Grundeken MJ, Kraak RP, Hassell ME, Arkenbout EK, Baan J Jr, Vis MM, Koch KT, Tijssen JG, Piek JJ, de Winter RJ, Henriques JP, Wykrzykowska JJ. Amsterdam Investigator-initiateD Absorb strategy all-comers trial (AIDA trial): a clinical evaluation comparing the efficacy and performance of ABSORB everolimus-eluting bioresorbable vascular scaffold strategy vs the XIENCE family (XIENCE PRIME or XIENCE Xpedition) everolimus-eluting coronary stent strategy in the treatment of coronary lesions in consecutive all-comers: rationale and study design. Am Heart J. 2014 Feb;167(2):133-40. doi: 10.1016/j.ahj.2013.09.017. Epub 2013 Oct 17. PMID 24439973
- [Derived] Kerkmeijer LSM, Renkens MPL, Tijssen RYG, Hofma SH, van der Schaaf RJ, Arkenbout EK, Weevers APJD, Garcia-Garcia HM, Kraak R, Piek JJ, Tijssen JGP, Henriques JPS, de Winter RJ, Wykrzykowska JJ. Long-term clinical outcomes of everolimus-eluting bioresorbable scaffolds versus everolimus-eluting stents: final five-year results of the AIDA randomised clinical trial. EuroIntervention. 2022 Mar 18;17(16):1340-1347. doi: 10.4244/EIJ-D-21-00419. PMID 34483094
- [Derived] Wykrzykowska JJ, Kraak RP, Hofma SH, van der Schaaf RJ, Arkenbout EK, IJsselmuiden AJ, Elias J, van Dongen IM, Tijssen RYG, Koch KT, Baan J Jr, Vis MM, de Winter RJ, Piek JJ, Tijssen JGP, Henriques JPS; AIDA Investigators. Bioresorbable Scaffolds versus Metallic Stents in Routine PCI. N Engl J Med. 2017 Jun 15;376(24):2319-2328. doi: 10.1056/NEJMoa1614954. Epub 2017 Mar 29. PMID 28402237